CLINICAL TRIAL: NCT00466219
Title: Ribavirin/Pegasys Treatment of Recurrent Hepatitis C After Liver Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SASL17
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Hepatitis C
Keywords: Presence of HCV RNA in serum; Absence of graft rejection; Recurrent hepatitis C after liver transplantation
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ribavirin
Drug: Pegylated interferon alpha2a

SUMMARY:
The aim of the study is to assess whether patients with recurrent hepatitis C after liver transplantation will benefit from a treatment with ribavirin/PEG-IFN-alpha combined treatment for 48 weeks.

DETAILED DESCRIPTION:
The aim of the study is to assess whether patients fulfilling the criteria as defined in section 3 will benefit from a treatment with ribavirin/PEG-a-IFN combined treatment. This study will be open to all patients with histologically documented hepatitis C recurring after LT, provided that all inclusion and exclusion criteria, as defined below, are met, and irrespectively of the pattern of response to a previous antiviral treatment (if any).

The benefit will be assessed in terms of biochemical (normalization of serum transaminases levels), virological (disappearance of HCV RNA from serum) and histological (amelioration of the histological signs of hepatitis) response. The presence of a sustained virological response, as defined below in section 6, will also be studied in relation to the early kinetics of serum HCV RNA, in keeping with recent data obtained in chronic hepatitis C patients, which suggest that an early rapid decrease of HCV viremia is associated with a durable response.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 year old patients, male or female, having undergone a LT for end-stage liver disease due to HCV
* patients presenting after LT with recurrent HCV infection, documented by presence of HCV RNA in serum, and recurrent hepatitis, diagnosed at histology; the liver biopsy upon which the diagnosis is established must have been performed within the 12 months prior to inclusion; the treatment cannot start within the 6 months following LT
* alpha fetoprotein value within normal limits obtained within 3 months before entry visit
* stable immunosuppressive regimen, defined as lack of any therapeutic measures aimed at preventing or treating graft rejection during the three months prior to antiviral therapy

Exclusion Criteria:

* participation in other clinical trial within 30 days of entry into this protocol
* patients retransplanted for rejection or for recurrent hepatitis C on the graft
* patients with a history of cardiovascular disease including but not limited to uncontrolled hypertension, angina pectoris, myocardial infarction, coronary artery surgery and congestive heart failure are excluded
* presence of HBsAg and/or HIV
* history of auto-immune disease, including auto-immune hepatitis
* alcohol consumption exceeding 40 grams per day
* acute rejection episode within the 3 months prior to inclusion, or current histological features possibly related to underlying rejection
* hepatocellular carcinoma
* unresolved biliary complication
* renal insufficiency (serum creatinine levels above 200 micromol/l)
* unconjugated bilirubin blood level > 100 micromol/l
* gammaglutamyl transferase > 20 times the upper limit of normal range
* prothrombin time below 60% of control (except in case of oral anti-coagulant therapy)
* neutrophil count less than 1,500/mm3
* platelet count less than 90,000/mm3
* hemoglobin below the lower limit of normal of the testing laboratory
* other organ or bone marrow transplantation
* current neoplasm and/or anti-tumor chemotherapy
* current hepatic arterial thrombosis
* pregnant or breast feeding women; child bearing potential women without adequate contraception throughout the course of therapy
* psychosis or anti-depressant therapy for uncontrolled clinical depression
* clinically significant retinal abnormalities
* thyroid dysfunction (abnormal TSH value with or without clinical symptoms)
* immunosuppressive therapy with OKT3 or any other anti-lymphocyte serum
* drug abuse (heroin, cocaine) or substitution therapy during the 12 months prior to inclusion
* history of ischemic cardiopathy
* interstitial pneumonitis
* previous auto-immune hemolysis and all causes of chronic hemolysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2002-05; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Biochemical (normalization of serum transaminases levels),
virological (disappearance of HCV RNA from serum)
and histological (amelioration of the histological signs of hepatitis) response.

SECONDARY OUTCOMES:
Correlation of the above outcome measures with early on-treatment HCV RNA dynamics (if applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Negro, MD, Principal Investigator — University Hospital, Geneva